CLINICAL TRIAL: NCT05872022
Title: Wegovy® (Semaglutide 2.4 mg) Pregnancy Registry Study: A Prospective Cohort Study to Investigate Safety Outcomes of Exposure to Wegovy During Pregnancy
Brief Title: A Study to Evaluate Safety of Exposure to Wegovy During Pregnancy
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-4937; U1111-1273-4336 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-04-26; First posted 2023-05-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants Exposed to Wegovy: Pregnant women who are exposed to Wegovy at any time during pregnancy for the treatment of obesity or overweight with at least one weight-related comorbid condition will be observed in this prospective observational study.
  Interventions: Other: No Intervention
- Participants Unexposed to Wegovy or Other GLP-1 RAs: Pregnant women who have overweight with at least one weight-related comorbid condition or who have obesity at conception and who are not exposed to Wegovy or other GLP-1 RAs at any time during pregnancy but who may be exposed to other products for weight management will be observed in this prospective observational study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study, therefore no intervention is used.

SUMMARY:
This is an observational, prospective Wegovy (semaglutide 2.4 milligram [mg]) Pregnancy Registry Study. The aim of this study is to compare the maternal, foetal, and infant outcomes of pregnant women who are exposed to Wegovy during pregnancy for the treatment of obesity or overweight with at least one weight-related comorbid condition with outcomes in an internal comparison cohort of pregnant women with obesity or overweight with at least one weight related comorbid condition at conception and who are not exposed to Wegovy or other glucagon-like peptide-1 receptor agonists (GLP-1 RAs) during pregnancy. Infant outcomes will be assessed throughout the infant's first year of life, with active data collection by the registry occurring at 4 and 12 months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities
* Female 15-50 years of age at the time of signing consent
* Currently or recently pregnant
* Resident of country included in the study
* Authorisation for her HCP(s) to provide data to the registry
* Exposed to Wegovy cohort: Exposure to at least one dose of Wegovy at any time during pregnancy for the treatment of obesity or overweight with at least one weight-related comorbid condition.
* Unexposed to Wegovy cohort: Have obesity or overweight with at least one weight related comorbid condition at conception

Exclusion Criteria:

* Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation
* Unexposed to Wegovy cohort: Exposure to Wegovy or other GLP-1 RA at any time during pregnancy

Ages: 15 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — This is a study of prenatal exposure to Wegovy in pregnant women.
Study Population: Pregnant participants exposed to Wegovy during pregnancy, and pregnant participants who were not exposed to Wegovy or other GLP-1 RAs at any time during pregnancy but who may be exposed to other products for weight management with obesity and overweight were to be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2032-10-31 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Infants with Major Congenital Malformation (MCM) | From date of conception (DOC) to pregnancy outcome for foetal losses or 12 months of infant age for live births
  Number of infants with MCM is defined as an abnormality of body structure or function that is present at birth; is of prenatal origin (that is, birth defect); has significant medical, social, or cosmetic consequences for the affected individual; and typically requires medical intervention.

SECONDARY OUTCOMES:
Number of Infants with Minor Congenital Malformation | From DOC to pregnancy outcome for foetal losses or 12 months of infant age for live births
  Number of infants with minor congenital malformation is defined as an anomaly or abnormality of body structure that is present at birth, is of prenatal origin (that is, birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual.
Number of Pregnant Participants With Pre-eclampsia | From 20 0/7 gestational weeks to 6 weeks
  Number of pregnant participants with pre-eclampsia is defined as pregnant participants with high blood pressure and signs of liver or kidney damage occurring at greater than (>) 20 gestational weeks through 6 weeks postpartum.
Number of Pregnant Participants With Eclampsia | From 20 0/7 gestational weeks to 6 weeks
  Eclampsia is defined as seizures or coma in a woman with pre-eclampsia during pregnancy through 6 weeks postpartum.
Number of Pregnant Participants Experiencing Spontaneous Abortion | From date of conception to 19 6/7 gestational weeks
  Number of pregnant participants experiencing spontaneous abortion is defined as an involuntary foetal loss or the expulsion of the products of conception occurring at less than (<) 20 gestational weeks.
Number of Pregnant Participants Experiencing Stillbirth | From 20 0/7 gestational weeks to pregnancy outcome (week 40)
  Number of pregnant participants experiencing still birth is defined by the American College of Obstetricians and Gynecologists (ACOG), an involuntary foetal loss occurring at greater than or equal to (>=)20 gestational weeks or, if gestational age is unknown, a foetus weighing >=350 gram.
Number of Pregnant Participants With Elective Termination | From date of conception to pregnancy outcome (week 40)
  Number of pregnant participants with elective termination is defined as a voluntary foetal loss or interruption of pregnancy that occurs for any reason, including but not limited to for the preservation of maternal health or due to foetal abnormalities.
Number of Pregnant Participants With Preterm Delivery | From date of conception to 37 gestational weeks (week 37)
  Preterm birth is defined as a live birth occurring at <37 gestational weeks.
Number of Infants Experiencing Small for Gestational Age (SGA) Birth | At delivery of live birth
  Number of infants experiencing small for gestational age is defined as weight at birth in <10th percentile for sex and gestational age using standard growth charts for full and preterm live born infants.
Number of Infants With Postnatal Growth Deficiency | At 4 and 12 months of infant age
  Number of infants with postnatal growth deficiency is defined as infants with weight, length, or head circumference in <10th percentile for sex and age using standard growth charts.
Number of infants with Developmental Delay | At 4 and 12 months of infant age
  Infant development delay is defined as infants with failure to achieve the developmental milestones for age, as defined by the Centers for Disease Control and Prevention (CDC).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834)., Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on NovoNordisk-trials.com
URL: http://novonordisk-trials.com